CLINICAL TRIAL: NCT03252561
Title: Ultrasound Guided Transversus Abdominis Plane (TAP) Block for Postoperative Analgesia After Laparoscopic Appendicectomy in Adults: A Double Blind Randomised Controlled Trial
Brief Title: TAP Block for Laparoscopic Appendicectomy in Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study no longer feasible
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sponsorship No. 249
Record Dates: First submitted 2015-04-20; First posted 2017-08-17 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Acute Appendicitis
Keywords: TAP block; Acute Appendicitis; Post-operative analgesia
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block (Experimental): Patients in this arm will receive ultrasound guided TAP bock with Bupivacaine 0.25% 20ml per side or to a maximum 1mg/kg per side and the skin puncture will be covered with a small plaster
  Interventions: Procedure: Ultrasound guided Transversus Abdominis Plane (TAP) bock
- Local anaesthetic infiltration (Active Comparator): Laparoscopic port sites will be infiltrated with a total of 20 mls 0.5% bupivacaine subcutaneously at the end of the procedure in the control group and plasters will be stuck on either side approximately where a skin puncture for tap block would be made.
  Interventions: Procedure: Local anaesthetic infiltration of laparoscopic port sites

INTERVENTIONS:
Procedure: Ultrasound guided Transversus Abdominis Plane (TAP) bock — Ultrasound guided TAP bock with Bupivacaine 0.25% 20ml per side or to a maximum 1mg/kg per side and the skin puncture will be covered with a small plaster
  Arms: TAP block
Procedure: Local anaesthetic infiltration of laparoscopic port sites — Laparoscopic port sites will be infiltrated with a total of 20 mls 0.5% bupivacaine subcutaneously at the end of the procedure in the control group and plasters will be stuck on either side approximately where a skin puncture for tap block would be made.
  Arms: Local anaesthetic infiltration

SUMMARY:
Laparoscopic (key-hole) appendicectomy is a minimally invasive procedure when compared to open large bowel resection, but is still associated with a significant amount of pain and discomfort. Analgesia is commonly provided by a multi-modal technique involving varying combinations of paracetamol, Non steroidal anti-inflammatory drugs (NSAIDs), regional analgesia and oral or parenteral opioids. Opioids are associated with an increased incidence of nausea, vomiting and sedation which can complicate post-operative recovery. Different techniques of intraoperative infiltration of local anaesthetic to control postoperative pain are also being used. Their perceived benefits are thought to relate to reduced opioid consumption and therefore reduced opioid side effects.

Transversus Abdominis Plane (TAP) block is a technique which numbs the nerves carrying pain sensation from the abdominal wall and provides effective and safe analgesia with minimal systemic side effects. Their perceived benefits are thought to relate to reduced opioid consumption and therefore reduced opioid side effects. The investigators believe ultrasound guided TAP blocks will reduce pain and morphine consumption with a resultant improved patient satisfaction, a reduction in post-operative nausea and vomiting and earlier hospital discharge.

The key research question the investigators are trying to answer is whether TAP block provide better pain relief than local anaesthetic infiltration of the laparoscopic port sites. Both techniques are currently being used in the investigator's hospital.

DETAILED DESCRIPTION:
Summary of Study Design: The study will be a double blind randomised controlled trial with patients undergoing laparoscopic appendicectomy randomly allocated into two groups. The study group will receive bilateral TAP blocks and the control group will receive local anaesthetic infiltration of the laparoscopic port sites

A double blind design was chosen to eliminate patient and observer bias in reporting of pain scores.

The presence of the control arm will ensure that any difference observed will be due to the effect of sensory nerve block due to the TAP block than due to the systemic effect of the injected local anaesthetic.

The null hypothesis will be that there is no difference between the groups in the amount of opioids consumed by the patients during 24 hours after the operation. The investigators chose this measurement as an objective but indirect measurement of efficacy of TAP block and pain relief thus received. Measurement of pain with various scoring methods are reliable only when concurrent reduction in consumption of pain killers are demonstrated.

Recruitment and randomisation:

All patients meeting the inclusion criteria will receive a patient information leaflet about the study during the procedure and investigators will gain informed consent during the procedure consultation. Investigators aim to recruit 288 patients with 144 patients in each group.

Informed consent will be taken the evening before, or on the morning of, surgery. Patients will then be randomly allocated into either the study group or a control group. Randomisation will occur by using computer generated random numbers using the block randomisation method. Group allocation will be kept in a consecutively numbered, opaque, sealed envelope in the controlled drugs cupboard in theatre-4/emergency theatre anaesthetic room of the John Radcliffe Hospital. Once the patient has consented, the anaesthetist will open the corresponding numbered envelope and perform bilateral TAP blocks after induction of general anaesthesia if the patient is in the study group. The surgeons will infiltrate the port sites with local anaesthetic at the end of the procedure if the patient is in the control group.

Blinding:

The study group will receive bilateral TAP blocks with 20mls 0.25% bupivacaine on each side and the skin punctures on either sides will be covered with a small plaster. Patients in the control group will receive subcutaneous infiltration of the laparoscopic port sites and specimen extraction site with equivalent amount bupivacaine at the end of the procedure and small plasters will be stuck on either flanks approximately where the skin punctures for TAP block will be made.

The assessor of pain scores and morphine doses (Recovery nurse, Ward Nursing Staff & SEU Foundation Doctor) and the patient will be blinded to group allocation.

Patient: Plasters will be stuck on flanks of all the patients, both study and control group, so that patient will not know if they have received TAP block.

Recovery nurse: During handover to recovery the anaesthetist and scrub nurse will not mention group allocation.

SEU Foundation Doctor: The foundation doctor who will be following up patients on the ward will not be present in the operating theatre, ensuring that they are blinded to the technique used.

The study duration will be from induction of anaesthesia until the patients are medically fit for discharge from hospital. No extra visits other than routinely required for the surgical procedure are expected.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to give informed consent for participation in the study
* Male or Female, aged 16 years or above
* Undergoing laparoscopic appendicectomy for a clinical diagnosis of appendicitis
* American Society of Anaesthetists physical status (ASA) 1-3

Exclusion Criteria:

* Opioid tolerance
* Chronic abdominal pain
* Allergy/Intolerance: Morphine, local anaesthetics, tramadol
* BMI (Body Mass Index) >35 Kg/M2
* Previous major abdominal surgery
* High likelihood of conversion of open procedure
* Patients unable to communicate in written and spoken English
* Weight less than 50 kg
* ASA > 3

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Opioid consumption in the first 12 hours after the operation | 12 hours
  The primary endpoint will be consumption of morphine or other opioids (including tramadol) in the first 12 hours after the operation. This will be recorded from the drug chart. Morphine equivalents include fentanyl, codeine and tramadol and will be converted into total morphine consumption using recognised conversion ratios.

SECONDARY OUTCOMES:
Numerical rating pain scores at emergence, 6, 12, 24 hours postoperatively | 24 hours after the operation
Time to first request for rescue analgesia | 24 hours after the operation
  The time will be calculated from the drug chart looking up when the first dose of rescue opioid was administered
Nausea score at emergence, 6, 12, 24 hours postoperatively | 24 hours after the operation
Total length of hospital stay | After the operation patients will be followed up till they are medically fit to be discharged from the hospital an expected length of 1-5 days
  Time will be calculated from the medical notes, when the decision that the patient is medically fit to be discharged was made
Opioid consumption at 24 hours | 24 hours after the operation
  Consumption of morphine or other opioids (including tramadol) in the first 24 hours after the operation. This will be recorded from the drug chart. Morphine equivalents include fentanyl, codeine and tramadol and will be converted into total morphine consumption using recognised conversion ratios

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silva, MBBS,MD,FRCS, Principal Investigator — Consultant Upper G Surgeon; Nicholas Crabtree, MBChB,FRCA, Principal Investigator — Consultant Anaesthetist
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

REFERENCES:
- [Background] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014
- [Background] Sandeman DJ, Bennett M, Dilley AV, Perczuk A, Lim S, Kelly KJ. Ultrasound-guided transversus abdominis plane blocks for laparoscopic appendicectomy in children: a prospective randomized trial. Br J Anaesth. 2011 Jun;106(6):882-6. doi: 10.1093/bja/aer069. Epub 2011 Apr 18. PMID 21504934
- [Background] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838